CLINICAL TRIAL: NCT05819593
Title: A Critical Analysis of Anaplastic Thyroid Clinical Trials: Perspectives From Patient Experiences
Brief Title: Evaluating Trends in Anaplastic Thyroid Cancer Patients' Clinical Study Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 80865259
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Anaplastic Thyroid Cancer
Keywords: anaplastic thyroid cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials can sometimes favor certain demographic groups. Additionally, there is limited research that delves into the factors that influence participation in clinical study, both positive and negative.

The goal is to identify the obstacles and challenges that prevent participation in anaplastic thyroid cancer clinical research, as well as the reasons for withdrawal or discontinuation.

Insights gained from this study will ultimately benefit those with anaplastic thyroid cancer who may be invited to participate in clinical research in the years to come.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with anaplastic thyroid cancer
* Willing to comply with all study related procedures and assessments
* Capable of giving signed informed consent, which includes compliance with requirements and restrictions listed in the informed consent form (ICF) and in the protocol

Exclusion Criteria:

* No documented diagnosis of anaplastic thyroid cancer
* Any serious and/or unstable pre-existing medical disorders
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anaplastic thyroid cancer who are actively considering participating in an observational clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of anaplastic thyroid cancer patients who decide to enroll in a clinical study | 3 months
Rate of anaplastic thyroid cancer patients who remain in a clinical study to completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Jundi M, Thakur S, Gubbi S, Klubo-Gwiezdzinska J. Novel Targeted Therapies for Metastatic Thyroid Cancer-A Comprehensive Review. Cancers (Basel). 2020 Jul 29;12(8):2104. doi: 10.3390/cancers12082104. PMID 32751138
- [Background] Saini S, Tulla K, Maker AV, Burman KD, Prabhakar BS. Therapeutic advances in anaplastic thyroid cancer: a current perspective. Mol Cancer. 2018 Oct 23;17(1):154. doi: 10.1186/s12943-018-0903-0. PMID 30352606
- [Background] Ljubas J, Ovesen T, Rusan M. A Systematic Review of Phase II Targeted Therapy Clinical Trials in Anaplastic Thyroid Cancer. Cancers (Basel). 2019 Jul 4;11(7):943. doi: 10.3390/cancers11070943. PMID 31277524

DOCUMENTS (1):
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT05819593/ICF_000.pdf